CLINICAL TRIAL: NCT05963334
Title: A Non-randomized Control Study Comparing Weekly Versus Every Three Weeks of Carboplatin Plus Paclitaxel in Patients With Advanced Epithelial Ovarian Cancer
Brief Title: Comparison of Weekly Versus Every Three Weeks of Carboplatin Plus Paclitaxel in Patients With Advanced Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Misr International University (Other)
Responsible Party: Principal Investigator, Omar Khaled Mohamed Abdel Monem Abo Hussein, Teaching and research assistant at the clinical pharmacy department, faculty of pharmacy, Misr International University, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PT 1491
Record Dates: First submitted 2023-07-10; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Advanced Epithelial Ovarian Cancer
Keywords: Carboplatin induced side effects; Patient safety; Acute and chronic kidney injury; Anemia, neutropenia and thrombocytopenia; Advanced epithelia ovarian cancer; Improved patient toleration; Patient counselling and education; Routine laboratory tests and tumor markers comparison; Additional biomarkers; Cystatin-C (Cys-C); Neutrophil gelatinase associated lipocalin (NGAL); Interleukin-18 (IL-18); Hepcidin (HEPC); Kidney injury marker-1 (KIM-1); Quality of life; Health related quality of life outcomes; Progression free survival; Palliative care; Chemotherapy, surgery and non-pharmacological treatment of ovarian cancer; Functional assessment of cancer therapy for ovarian cancer (FACT-O); Functional assessment of cancer therapy/gynecologic oncology group/neurotoxicity (FACT-GOG/NTX)
MeSH Terms: conditions — Anemia; Neutropenia; Thrombocytopenia | interventions — CP protocol

STUDY DESIGN:
Intervention Model Description: prospective open-label non-randomized control study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weekly dose of carboplatin / paclitaxel (n=21) (Experimental): Patients in this group received the weekly dose regimen, where the dose of carboplatin administered intravenously once/week was calculated using the Calvert equation to yield an area under the curve (AUC) = 2
  Interventions: Drug: Carboplatin/paclitaxel
- 3-Week collective dense dose of carboplatin / paclitaxel (n=28) (Active Comparator): Patients in this group received the three-week collective dose regimen, where the dose of carboplatin was administered intravenously once on day 1/ every three weeks (21 days) and was calculated using the Calvert equation to yield an AUC = 6
  Interventions: Drug: Carboplatin/paclitaxel

INTERVENTIONS:
Drug: Carboplatin/paclitaxel — Weekly dose versus every three weeks dense dose of carboplatin/paclitaxel regimen in advanced epithelial ovarian cancer.

SUMMARY:
The aim of the current study is to compare weekly versus three-week collective of carboplatin/paclitaxel in advanced epithelial ovarian cancer. The author's hypothesis was to study and correlate routine laboratory tests, clinical biomarkers and quality of life questionnaires between weekly and three-week standard carboplatin regimens in order to reveal any possible superiority for the weekly study arm.

DETAILED DESCRIPTION:
Ovarian cancer as the fifth leading cause of death in women worldwide. Since most women suffer asymptomatic manifestations or nonspecific symptoms, subsequent diagnosis is very tricky and late most of the time. Carboplatin/paclitaxel has been among the first line options for treatment of ovarian cancer for decades however, account for a great of deal of adverse effects affecting patient safety. These side effects are dose related whereas, dose of carboplatin is calculated individually for each patient using the Calvert equation focusing on renal functions at baseline. Carboplatin adverse effects are believed to mainly affect the kidneys, hematological system and may cause neurotoxicity thus, exhibit quality of life deteriorations.

The study purpose was to investigate a triple correlation between 3 different aspects comparing the weekly dose versus the three-week dense dose of carboplatin/paclitaxel in treating advanced epithelial ovarian cancer.

Points of comparison:

1. Routine laboratory parameters in an attempt to identify the possible adverse effects accounted to each regimen focusing on hematological, renal, hepatic, and tumor marker panels.
2. Additional biomarkers including cystatin-C, neutrophil gelatinase associated lipocalin, hepcidin, kidney injury marker-1 and interleukin-18 assessing the probable incidence of acute kidney injury and anemia.
3. Quality of life analyzed by comparing functional assessment of cancer therapy-ovarian and functional assessment of cancer therapy/gynecologic oncology group-neurotoxicity surveys between both groups.

The study encouraged the patient right to be involved and consent to the assigned protocol

The correlation between all three aspects studied as of routine lab work, toxicity biomarkers and quality of life besides the economic burden aim to provide a decent patient tailored treatment regimen balancing efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Cancer stage according to the International Federation of Gynecology and Obstetrics (FIGO) classification subdivided into the following categories; (I A, B, and C), II (A and B) III (A, B and C) and (IVA and B). Stage I: (tumor limited to the uterus (confined to the organ of origin) and subdivided into IA: below 5cm, IB : above 5 cm.

Stage II: Tumor extends beyond the uterus within the pelvis (invasion of surrounding organs) subdivided into IIA: adnexal involvement, IIB: involvement of other pelvic tissue.

Stage III: Tumor invades abdominal tissue (spread to nodes or tissue within the pelvis), subdivided into: IIIA: one site; IIIB: more than one site; IIIC: metastasis to the pelvic and/or para-aortic lymph node.

Stage IV: Tumor invades external organs to the uterus subdivided into IVA: tumor invading the bladder and/or rectum while IVB: distant metastasis(es).

-Indication for chemotherapy and life expectancy of at least 3 months Performance status is above and equal to 3 according to the Eastern Cooperative Oncology Group (ECOG).

Exclusion Criteria:

* Heart disease (congestive heart failure, myocardial infarction within 6 months from study entry, atrioventricular block of any grade, severe arrhythmias)
* Neutrophils (ANC) < 2000 x mm3, platelets (PLT) < 100,000 x mm3
* Inadequate renal function {creatinine (SCr) ≥1.5 x normal values} or liver function (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 1.5 x normal values).

Discontinuation criteria:

* Present or suspected hemorrhagic syndromes
* Inability to comply with protocol and follow-up
* Inability to access the study site for clinical visits
* Refusal of informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Epithelial ovarian cancer patients
Enrollment: 49 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Routine blood work and tumor markers | 6 cycles for each patient with a total of126 days
  Quantitative continuous parameter assay of blood samples to measure hemoglobin gram/deciliter, total leukocyte count, platelets, neutrophils all in (number/unit liter), serum creatinine, blood urea nitrogen, uric acid, serum calcium in (milligram/deciliter), alanine aminotransferase, aspartate aminotransferase in (unit liter), albumin (gram liter), carcinoembryonic antigen (nano-gram milliliter), and cancer antigen-125 (unit milliliter)
  This was cross-referenced against the universal laboratory values to identify the degree of anemia, neutropenia, thrombocytopenia, calcium deficiency, kidney injury, liver toxicity, and tumor progression comparing pre-and post-treatment results for patients on each regimen separately and also compare post-treatment between the two regimens by end of treatment (weekly dose of carboplatin group and 3-week collective dense dose carboplatin regimens).
Additional kidney and anemia biomarkers | 6 cycles for each patient with a total of126 days
  Cystatin-C ng/mL, Neutrophil gelatinase-associated lipocalin ng/mL, Interleukin-18 pg/mL, Kidney injury marker-1 ng/mL, and Hepcidin pg/mL
  Acute kidney injury to the glomerular capsule and proximal tubule was assessed by the increase in Cys-C, NGAL, KIM-1, and IL-18 Anemia and diminished renal clearance resembling kidney injury were measured by increased levels of HEPC
  Pre-and post-treatment concentrations were compared for patients on each carboplatin regimen & post-treatment concentration by the end of treatment between weekly and collective 3-week dense dose
  * Biomarkers were measured using ELISA reader
  * Absorbance was converted to serum concentration using the standard curve for each biomarker constructed using the readings for standard serial dilutions
  * Concentrations were used to compare regimens and outline the carboplatin dosing schedule with the least margin of toxicity
  (Higher marker levels outline greater toxicity)
Improved quality of life | 6 cycles for each patient with a total of126 days
  Functional assessment of cancer therapy-ovarian (FACT-O) & functional assessment of cancer therapy/Gynecologic Oncology Group neurotoxicity (FACT-GOG-NTX)
  A 5-point Likert-type scale ranging from 0 (not at all) to 4 (very much). FACIT organization developed questions into 5 compartments: {Personal (PWB), Emotional (EWB), Social (SWB), Functional (FWB), Ovarian cancer (OC) & Neurotoxicity (NTX))
  Hard copies, consume 10-15 mins to fill, patients documented their responses, guideline reverse calculation & trial outcome indices analyzed
  Compared at baseline, post-treatment by the end of therapy for each group individually & post-treatment between both carboplatin regimens FACT-G total score = PWB + EWB + SWB + FWB FACT-O total score = PWB + EWB + SWB + FWB + OC FACT/GOG-Ntx total score = PWB + EWB + SWB + FWB + NTX FACT-O Trial Outcome Index (TOI) = PWB + FWB + OC FACT/GOG-Ntx Trial Outcome Index (TOI) = PWB + FWB + NTX
  High scores = enhanced QOL, low scores = poor QOL

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmacology and toxicology department, Faculty of Pharmacy, Cairo University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Study findings, Experimental module, Ethical approval, Patient consent, Inclusion criterion, Exclusion criteria, Baseline characteristics.